CLINICAL TRIAL: NCT04614246
Title: A Randomized, Double-blind, Open for Active Comparator, Parallel-group, Multicenter Phase 2b Study to Assess the Efficacy and Safety of Three Different Doses of P2X3 Antagonist (BAY1817080) Versus Placebo and Elagolix 150 mg in Women With Symptomatic Endometriosis
Brief Title: Study to Gather Information How Well Three Different Doses of BAY1817080 Given Twice Daily Over 12 Weeks Work in Comparison to an Inactive Pill (Placebo) and Elagolix in Women Suffering From Pain Related to a Condition Where the Tissue That Usually Grows Inside the Womb Grows Outside of the Womb
Acronym: SCHUMANN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by Sponsor
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20584; 2020-003131-16 (EudraCT Number)
Record Dates: First submitted 2020-11-02; First posted 2020-11-03 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — elagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind to placebo and open-label for active comparator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BAY1817080 150 mg (Experimental): Participants will receive 150 mg of BAY1817080 twice daily over a 12-week intervention period
  Interventions: Drug: BAY1817080
- BAY1817080 75 mg (Experimental): Participants will receive 75 mg of BAY1817080 twice daily over a 12-week intervention period
  Interventions: Drug: BAY1817080
- BAY1817080 25 mg (Experimental): Participants will receive 25 mg of BAY1817080 twice daily over a 12-week intervention period
  Interventions: Drug: BAY1817080
- Elagolix (Active Comparator): Participants will receive 150 mg of Elagolix once daily over a 12-week intervention period
  Interventions: Drug: Elagolix
- Placebo (Placebo Comparator): Participants will receive placebo matching BAY1817080 twice daily over a 12-week intervention period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY1817080 — Tablet, oral administration
  Arms: BAY1817080 150 mg; BAY1817080 25 mg; BAY1817080 75 mg
Drug: Elagolix — Tablet, oral administration
  Arms: Elagolix
Drug: Placebo — Tablet, oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess safety and efficacy of BAY 1817080 compared to elagolix and placebo in women with symptomatic endometriosis. Study details include:

* Study duration: 155 up to 285 days
* Treatment duration: 84 days
* Visit frequency: 3 laboratory every 2 weeks for participants on BAY 1817080 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age at the time of signing the informed consent
* Visually-confirmed endometriosis: detection of endometriotic lesions during laparoscopy or laparotomy (with or without pathological diagnosis) within 10 years but no less than 8 weeks from Visit 1a (surgically diagnosed endometriosis). For Japan only and limited to no more than half of all randomized Japanese participants: the diagnosis can be based on previous imaging (i.e. endometriosis lesion detected by ultrasound or MRI). If the participant was diagnosed by ultrasound, the lesion must be visualized again by ultrasound at the screening visit. If the participant was diagnosed by MRI, the diagnosis must have been made within 12 months before Visit 1a (clinically diagnosed endometriosis).
* Both sub-criteria regarding pain symptoms must be fulfilled:

  * At Visit 1a, participant presents self-reported moderate to severe pain which - based on the judgement of the investigator - carries a reasonable likelihood to translate into a severity of pain symptoms sufficient to fulfil the eligibility criterion and be caused by endometriosis, and
  * During the screening period at least 24 daily ESD entries during the 28 consecutive days starting on the first day with menstrual bleeding at or after Visit 1a and entries in the ESD item 1a ('worst pain' on the daily numerical rating scale) sum up to 98 or more.
* Willingness to use standardized rescue pain medications for EAPP (i.e. ibuprofen, acetaminophen and tramadol) and not use any prophylactic pain medication, according to investigator's instruction
* Ability to swallow the study intervention, i.e., the different kinds of tablets, as complete units
* Good general health (except for findings related to endometriosis) as proven by medical history, physical and gynecological examinations and laboratory test results
* Normal or clinically insignificant cervical cytology not requiring further follow-up:

  * A cervical cytology sample has to be obtained during screening, or
  * A documented normal result has to be available from cervical cytology conducted within 12 months prior to Visit 1a.
  * Human papilloma virus (HPV) testing in participants with atypical squamous cells of unknown significance (ASCUS) will be used as an adjunctive test automatically. Participants with ASCUS can be included if they are negative for high-risk HPV strains.

Exclusion Criteria:

* Current pregnancy or less than 3 months since delivery, abortion or stop of lactation before Visit 1a
* Hypersensitivity to any ingredient of the study intervention and/or the standardized rescue medications
* Known osteoporosis
* History of a low trauma fracture
* Contraindications for elagolix or the standardized rescue medications
* Current malignancy or history of cancer (exception: basal cell or squamous cell carcinoma of the skin) within the last 5 years prior to Visit 1a
* Any other diseases or conditions that according to the investigator can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study intervention (e.g. extremely low body weight, chronic bowel disease, Crohn's disease and ulcerative colitis)
* Menopause or signs of menopausal transition, such as absence of regular menstrual cycles based on investigator's judgment (absence of information regarding menstrual bleeding pattern e.g. due to long term use of hormonal contraception is not an exclusion criterion)
* Any disease or condition that may worsen during the study period according to the assessment and opinion of the investigator
* Abnormal uterine bleeding in terms of regularity or heaviness (with the exception of heavy menstrual bleeding that does not require treatment)
* Any findings that require further diagnostic procedures to avoid harm to the participant (e.g. ovarian tumors of uncertain origin or pelvic masses of unclear etiology)
* Any serious or unstable diseases or medical conditions, including psychiatric disorders, that might interfere with the conduct of the study or the interpretation of the result, including for example:

  * history of hysterectomy and/or bilateral oophorectomy
  * any conditions considered to contribute significantly to pelvic pain by the investigator, e.g. fibromyalgia, uterine fibroids, irritable bowel syndrome or other bowel disorders
  * any other underlying diseases requiring regular use of pain medication (e.g. migraine)
  * history of or current anxiety or depression unless stable with or without medical treatment ≥ 6 months before Visit 1a
* Major surgery scheduled during the study period
* Non-responsiveness of EAPP to earlier treatment with GnRH-agonists or GnRH-antagonists, based on the judgement of the investigator
* SARS-CoV-2- positive virus RNA test within 4 weeks prior to Visit 1a reported by participant, regardless of whether the participant had symptoms
* History of COVID-19 infection with persistent/ongoing symptoms
* Contact with SARS-CoV-2- positive or COVID-19 patient within the last 4 weeks prior to Visit 1a
* Intake of medication prohibited due to potential drug-drug interaction
* Use of other treatments that might interfere with the conduct of the study or the interpretation of the results, including:

  * hormonal medications
  * other treatments intended for endometriosis/pelvic pain during participation in the study, including the use of herbal products or traditional Chinese medicine for symptom relief, with the exception of the standardized rescue pain medications
* Simultaneous participation in another clinical trial with investigational medicinal product(s). Participation in another trial 3 months prior to Visit 1a that might have an impact on the study objectives, at the discretion of the investigator
* Previous assignment to study intervention (randomization) in this study (allowing previously randomized participants to be re-included into the study may lead to bias)
* Laboratory values outside the inclusion range (specified in the laboratory manual) and considered clinically relevant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (144):
- United States (46):
  - Accel Research Sites - Cahaba Medical Care, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mobile Ob-Gyn, PC, Mobile, Alabama
  - Precision Trials, AZ, LLC, Phoenix, Arizona
  - Diagnamics, Inc., Encinitas, California
  - West Coast OB/GYN Associates, San Diego, California
  - Advanced Women's Health Institute, Greenwood Village, Colorado
  - Office of Dr. James A. Simon, MD, Washington D.C., District of Columbia
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Alliance for Multispecialty Research, LLC - Fort Meyers, Fort Myers, Florida
  - Suncoast Clinical Research Center, Inc., New Port Richey, Florida
  - A Premier Medical Research of Florida, LLC, Orange City, Florida
  - Physician Care Clinical Research, Sarasota, Florida
  - Medisense, Inc., Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Paramount Research Solutions-College Park, College Park, Georgia
  - Journey Medical Research, Snellville, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Southern Clinical Research Associates LLC, Metairie, Louisiana
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Wayne State University Physicians Group, Detroit, Michigan
  - Essential Women's Health Associates, Las Vegas, Nevada
  - Bosque Womens Care, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Carolina Women's Research & Wellness Center, Durham, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Clinical Inquest Center, Ltd., Beavercreek, Ohio
  - Aventiv Research - Dublin, Dublin, Ohio
  - Centricity Research formerly Aventiv - Dublin, Dublin, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - University Hospitals Landerbrook Health Center, Mayfield Heights, Ohio
  - Palmetto Clinical Research, Summerville, South Carolina
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Medical Research Center of Memphis, LLC, Memphis, Tennessee
  - International Clinical Research-Tennessee LLC., Murfreesboro, Tennessee
  - Discovery Clinical Trials - Dallas, Dallas, Texas
  - UT Health Women's Research Center at Memorial City, Houston, Texas
  - Biopharma Informatic, Inc., Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Advances in Health, Pearland, Texas
  - Tidewater Clinical Research, Inc., Norfolk, Virginia
  - Eastern Virginia Medical School | OB/GYN Clinical Research Center, Norfolk, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Physicians For Women, North Chesterfield, Virginia
  - Seattle Clinical Research Center, Seattle, Washington
- Austria (2):
  - Medizinische Universität Graz, Graz, Styria
  - Universitätsklinikum AKH Wien, Vienna
- Belgium (4):
  - AZ Jan Palfijn Gent, Ghent, Oost-Vlaanderen
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Gent, Ghent
- Bulgaria (5):
  - MC Asklepii OOD, Dupnitsa
  - Spec. Hospital for Active Treatment of Oncological Diseases, Sofia
  - Medical Center Panaceya, Sofia
  - MHAT Niamed, Stara Zagora
  - SHOGAT Prof Dimitar Stamatov, Varna
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - The Ottawa Hospital | The Ottawa Hospital Research Institute - Neurology - Ottawa Stroke Program, Ottawa, Ontario
  - Clinique OVO, Montreal, Quebec
  - Alpha Recherche Clinique LB9, Québec
- China (7):
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Wuhan Tongji Reproductive Medicine Hospital, Wuhan, Hubei
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Beijing Obstetrics and Gynecology Hospital,Capital Med.Uni., Beijing
  - Peking University First Hospital, Beijing
- Czechia (9):
  - Fakultni nemocnice Brno, Brno
  - Gynekologie Meda s.r.o. - Lidicka, Brno-střed
  - GYN-MIKA s.r.o., České Budějovice
  - GynCare MUDr. Michael Svec s.r.o., Pilsen
  - Centrum gynekologicke rehabilitace, Písek
  - GYNERA, Prague
  - Gynekologie Studentsky dum s.r.o., Prague
  - Fakultní nemocnice Bulovka, Prague
  - Dr. Smrhova-Kovacs, Tábor
- Estonia (2):
  - Parnu Hospital, Pärnu
  - Clinic Elite, Tartu
- Finland (2):
  - HUS / Naistenklinikka, Helsinki
  - Lääkärikeskus Gyneko, Oulu
- Germany (5):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - emovis GmbH, Berlin
  - Charité - Campus Virchow-Klinikum (CVK), Berlin
- Greece (2):
  - ARETAIEION University Hospital, Athens
  - University General Hospital of Patras | Univ Obs & Gynae Cli, Pátrai
- Hungary (2):
  - Cortex Study Center, Budapest
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- Italy (6):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - ASST Sette Laghi, Varese, Lombardy
  - A.O.U. Careggi, Florence, Tuscany
  - A.O.U.I. Verona, Verona, Veneto
- Japan (20):
  - Aiiku Ladies Clinic, Funabashi, Chiba
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu, Chiba
  - Sou Clinic, Yotsukaidō, Chiba
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Social Medical Corporation Tokeidai Memorial Hospital, Sapporo, Hokkaido
  - Nishikawa Women's Health Clinic, Sapporo, Hokkaido
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Fujisawa City Hospital, Fujisawa, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Kurashiki Medical Clinic, Kurashiki, Okayama-ken
  - Suita Tokushukai Hospital, Suita, Osaka
  - Omi Medical Center, Kusatsu, Shiga
  - Kashiwazaki ladies clinic, Saitama, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Toyama Rosai Hospital, Uozu, Toyama
  - JCHO Tokuyama Central Hospital, Shūnan, Yamaguchi
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Saiseikai Nagasaki Hospital, Nagasaki
  - Nagasaki University Hospital, Nagasaki
- Latvia (4):
  - Latvian Maritime Medicine Center, Riga
  - Vitols and Vitols Ltd, Riga
  - I.Vasaraudzes Private Practice, Riga
  - I.Dinsbergas Physician Practice, Riga
- Lithuania (3):
  - JSC Seimos gydytojas family medical center, Vilnius
  - V. Jonaitienes private gynecology clinic, Vilnius
  - JSC Gyvenk Silciau Medical Center Maxmeda, Vilnius
- Norway (3):
  - Kirkeparken Spesialistpraksis, Fredrikstad
  - Oslo Universitetssykehus HF, Ullevål, Oslo
  - Sykehuset i Vestfold HF, Tønsberg, Tønsberg
- Poland (11):
  - Gabinet Ginekologiczny Janusz Tomaszewski, Bialystok
  - MICS Centrum Medyczne Torun, Bydgoszcz
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - NZOZ MEDEM Wilk Sp. j., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Prywatny Gabinet Lekarski Ginekologia, Poloznictwo i Ultr., Lodz
  - Specjalistyczny Gabinet Ginekologiczno-Polozniczy, Lublin
  - NZOZ NOVITA, Specjalistyczne Gabinety Lekarskie S.C, Lublin
  - VitroLive Sp. z o.o., Szczecin
  - MTZ Clinical Research Sp z o.o., Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
- Slovakia (3):
  - ULMUS, s r.o., Hlohovec
  - GA Lucenec s.r.o, Lučenec
  - Virina sano, s.r.o. Gynekologicko porodnicka ambulancia, Veľký Krtíš
- Spain (4):
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital de la Santa Creu i de Sant Pau | Ginecologia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Parke S, Gude K, Roth K, Messina F. Efficacy and safety of eliapixant in endometriosis-associated pelvic pain: the randomized, placebo-controlled phase 2b SCHUMANN study. BMC Womens Health. 2024 Jun 19;24(1):353. doi: 10.1186/s12905-024-03188-8. PMID 38890641
- [Derived] Fletcher MC. Selectivity of the P2X3 receptor antagonist Eliapixant, and its potential use in the treatment of endometriosis. Purinergic Signal. 2022 Mar;18(1):1-3. doi: 10.1007/s11302-021-09831-5. Epub 2022 Jan 3. No abstract available. PMID 34978027
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multinational study was conducted between 29 JAN 2021 First Patient First Visit (FPFV) and 03 MAY 2022 Last Patient Last Visit (LPLV) in 20 countries/regions: Austria, Belgium, Bulgaria, Canada, China, Czech Republic, Estonia, Finland , Germany, Greece, Hungary, Italy, Japan, Lithuania, Latvia, Norway, Poland, Slovakia, Spain, United States
Pre-assignment Details: A total of 215 participants were randomized to 5 treatment arms (44 to eliapixant, 44 to eliapixant, 43 to eliapixant, 43 to placebo, and 41 to Elagolix).
Groups:
- Eliapixant (BAY1817080) 25 mg: 25mg eliapixant twice daily for 12 weeks
- Eliapixant (BAY1817080) 75 mg: 75mg eliapixant twice daily for 12 weeks
- Eliapixant (BAY1817080) 150 mg: 150mg eliapixant twice daily for 12 weeks
- Placebo: Placebo for eliapixant twice daily for 12 weeks
- Elagolix 150mg: 150mg Elagolix once daily for 12 weeks
Period: Overall Study
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo | Elagolix 150mg
Started | 44 | 44 | 43 | 43 | 41
Valid for Safety Analysis Set (SAF) | 39 | 38 | 38 | 37 | 38
Completed | 28 | 22 | 22 | 24 | 24
Not Completed | 16 | 22 | 21 | 19 | 17
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 3
Not completed — Other reason | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 4 | 3 | 4
Not completed — Physician Decision | 0 | 2 | 1 | 0 | 0
Not completed — Study terminated by sponsor | 10 | 15 | 12 | 13 | 9
Not completed — Pregnancy | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) includes all 215 participants who were randomized to 5 treatment arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo | Elagolix 150mg | Total
Number analyzed (Participants) | 44 | 44 | 43 | 43 | 41 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 43 | 43 | 41 | 215
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 43 | 43 | 41 | 215
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 31 | 30 | 29 | 39 | 160
  Black or african american | 0 | 1 | 2 | 2 | 0 | 5
  Asian | 13 | 12 | 11 | 12 | 0 | 48
  Not reported | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Mean Worst Endometriosis Associated Pelvic Pain (EAPP), Primary Per Protocol Set (pPPS)
Description: The worst EAPP was measured daily on the 0-10 Numerical Rating Scale (NRS) by item 1 of the Endometriosis Symptom Diary (ESD). In question 1, participants were asked to rate the pain in the target area during the past 24 hours, where 0= no pain and 10= worst imaginable pain and responses were recorded in ESD. The absolute change in mean worst EAPP was from baseline (last 28 days before the first intake of study drug) to end of intervention (last 28 days ending with the last intake of study drug planned on Day 84 [+3]). The time frame of 28 days captures a menstrual cycle on average.
Time Frame: change from baseline to week 12
Population: The Elagolix arm was not included in the primary per protocol set (pPPS) simply because it's not part of the primary objective which was "to assess the dose-response relationship and demonstrate efficacy of BAY 1817080 compared to placebo in women with symptomatic endometriosis".
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Eliapixant (BAY1817080) 25 mg: Eliapixant 25 mg BID
- Eliapixant (BAY1817080) 75 mg: Eliapixant 75 mg BID
- Eliapixant (BAY1817080) 150 mg: 50 mg Eliapixant BID
- Placebo: Placebo for Eliapixant BID
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo
Number analyzed (Participants) | 31 | 31 | 31 | 30
units on a scale
  Baseline | 6.40 (1.66) | 6.13 (1.77) | 6.95 (1.38) | 6.14 (1.96)
  Week 12: number analyzed (Participants) | 24 | 22 | 20 | 26
  Week 12 | 4.57 (2.10) | 4.15 (2.49) | 5.15 (2.42) | 4.29 (1.71)
  Week 12: Change from Baseline: number analyzed (Participants) | 24 | 22 | 20 | 26
  Week 12: Change from Baseline | -1.56 (1.35) | -2.12 (2.66) | -1.88 (2.03) | -1.89 (1.91)
Statistical Analysis 1: Comparison: Eliapixant (BAY1817080) 25 mg; 80% confidence interval (CI) for change in mean worst EAPP from baseline to Week 12; Test type: Other; Mixed Models Analysis; LS-Mean = -1.63, 80% CI 2-sided [-2.13 to -1.14], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Eliapixant (BAY1817080) 75 mg; 80% confidence interval (CI) for change in mean worst EAPP from baseline to Week 12; Test type: Other; Mixed Models Analysis; LS-Mean = -2.13, 80% CI 2-sided [-2.66 to -1.61], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: Eliapixant (BAY1817080) 150 mg; 80% confidence interval (CI) for change in mean worst EAPP from baseline to Week 12; Test type: Other; Mixed Models Analysis; LS-Mean = -1.96, 80% CI 2-sided [-2.48 to -1.43], Standard Error of Mean 0.41
Statistical Analysis 4: Comparison: Placebo; 80% confidence interval (CI) for change in mean worst EAPP from baseline to Week 12; Test type: Other; Mixed Models Analysis; LS-Mean = -1.94, 80% CI 2-sided [-2.44 to -1.45], Standard Error of Mean 0.38

2. Secondary Outcome: Least Squares Mean (SE) Changes in Worst EAPP From Baseline to Week 12, Per Protocol Set
Description: as for outcome 1
Time Frame: change from baseline to week 12
Population: Per protocol set (PPS): includes 183 participants, which is 85.1% of the FAS population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Elagolix 150 mg: Elagolix 150 mg OD
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 37 | 37 | 36 | 36 | 37
units on a scale | -1.60 (0.40) | -2.07 (0.42) | -1.97 (0.42) | -1.89 (0.40) | -2.69 (0.41)
Statistical Analysis 1: Comparison: Eliapixant (BAY1817080) 25 mg vs Placebo; Difference of least square-mean (95% Confidence Interval, CI) - Eliapixant arms vs Placebo arm (pairwise comparison) - change in mean worst EAPP from baseline to Week 12 - pPPS; Test type: Other — mixed model repeated measures; Difference of least square-mean = 0.29, 95% CI 2-sided [-0.77 to 1.35], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: Eliapixant (BAY1817080) 75 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — mixed model repeated measures (MMRM); Difference of least square-mean = -0.18, 95% CI 2-sided [-1.27 to 0.91], Standard Error of Mean 0.55
Statistical Analysis 3: Comparison: Eliapixant (BAY1817080) 25 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — mixed model repeated measures (MMRM); Difference of least square-mean = -0.08, 98% CI 2-sided [-1.17 to 1.02], Standard Error of Mean 0.56
Statistical Analysis 4: Comparison: Eliapixant (BAY1817080) 25 mg vs Placebo; Difference of least square-mean (80% Confidence Interval, CI) - Eliapixant arms vs Placebo arm (pairwise comparison) - change in mean worst EAPP from baseline to Week 12 - pPPS; Test type: Other — mixed model repeated measures (MMRM); Difference of least square-mean = 0.29, 80% CI 2-sided [-0.4 to 0.98], Standard Error of Mean 0.54
Statistical Analysis 5: Comparison: Eliapixant (BAY1817080) 75 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Other — mixed model repeated measures (MMRM); Difference of least square-mean = -0.18, 80% CI 2-sided [-0.89 to 0.53], Standard Error of Mean 0.55
Statistical Analysis 6: Comparison: Eliapixant (BAY1817080) 150 mg vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Other — mixed model repeated measures (MMRM); Difference of least square-mean = -0.08, 80% CI 2-sided [-0.79 to 0.64], Standard Error of Mean 0.56

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: A treatment-emergent AE (TEAE) was defined as any event arising or worsening after the start of study drug administration until 14 days after the last study medication intake.
Time Frame: up to 14 days after the last study medication intake
Population: Safety analysis set (SAF) includes 190 participants (88.4%) since 25 participants (11.6%) did not receive any study intervention and was excluded from SAF.
Measure: Number; unit: Participants
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo | Elagolix 150 mg
Number analyzed (Participants) | 39 | 38 | 38 | 37 | 38
Participants
  Any TEAE | 23 | 21 | 29 | 27 | 28
  Any drug related TEAE | 4 | 6 | 10 | 10 | 13
  Any serious TEAE | 0 | 2 | 2 | 1 | 1
  Any drug related serious TEAE | 0 | 0 | 1 | 0 | 1
  Any TEAE with outcome death | 0 | 0 | 0 | 0 | 0
  Any TEAE resulting in permanent discontinuation of studly drug | 0 | 1 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 14 days after the last study medication intake with an average of 14 weeks. While for the all-cause mortality that occurred at any time during the study before the last contact, up to 285 days.
Description: A treatment-emergent AE (TEAE) was defined as any event arising or worsening after the start of study drug administration until 14 days after the last study medication intake.
Groups:
- Eliapixant (BAY1817080) 25 mg: 25 mg Eliapixant twice daily for 12 weeks
- Eliapixant (BAY1817080) 75 mg; Eliapixant (BAY1817080) 150 mg: 75 mg Eliapixant twice daily for 12 weeks
- Placebo: Placebo for 12 weeks
- 150 mg Elagolix: 150 mg Elagolix once daily for 12 weeks
Arm/Group | Eliapixant (BAY1817080) 25 mg | Eliapixant (BAY1817080) 75 mg | Eliapixant (BAY1817080) 150 mg | Placebo | 150 mg Elagolix
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38 | 0/38 | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 2/38 | 2/38 | 1/37 | 1/38
Other Adverse Events (participants affected / at risk) | 23/39 | 20/38 | 29/38 | 27/37 | 28/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliapixant (BAY1817080) 25 mg (N=39) | Eliapixant (BAY1817080) 75 mg (N=38) | Eliapixant (BAY1817080) 150 mg (N=38) | Placebo (N=37) | 150 mg Elagolix (N=38)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eliapixant (BAY1817080) 25 mg (N=39) | Eliapixant (BAY1817080) 75 mg (N=38) | Eliapixant (BAY1817080) 150 mg (N=38) | Placebo (N=37) | 150 mg Elagolix (N=38)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear swelling (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (6) | 1 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 4 (6) | 0 (0) | 4 (7) | 0 (0)
Vaccination site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Immune system disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Carbuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 5 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Blood glucose abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Full blood count abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coagulation test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (15) | 7 (11) | 6 (9) | 9 (17) | 8 (15)
Hypogeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Psychogenic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT04614246/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04614246/SAP_001.pdf